CLINICAL TRIAL: NCT00783744
Title: 28-week, Open, Randomized, Multinational, Multicenter Clinical Trial to Compare Efficacy and Safety of Combination Therapy of Glimepiride Plus Metformin Plus HOE901 Insulin Analogue Versus a Two-injection Conventional Therapy With Premixed Insulin NPH 30/70 Bid in Type 2 Diabetes Mellitus Patients Poorly Controlled With Oral Antidiabetic Drug Treatment.
Brief Title: Insulin Glargine Combination Therapies in Type II Diabetics
Acronym: LAPTOP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4027
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; glimepiride; Metformin

ARMS (2):
- 1 (Experimental): Insulin Glargine + Glimepiride + Metformin
  Interventions: Drug: Insulin Glargine; Drug: Glimepiride; Drug: Metformin
- 2 (Active Comparator): Insulin monotherapy with premixed insulin NPH 30/70
  Interventions: Drug: Insulin monotherapy with premixed insulin NPH 30/70

INTERVENTIONS:
Drug: Insulin Glargine — In the morning to target FBG ≤ 100 mg/dl
  Arms: 1
Drug: Glimepiride — Glimepiride 3 or 4 mg
  Arms: 1
Drug: Metformin — At least 850 mg od
  Arms: 1
Drug: Insulin monotherapy with premixed insulin NPH 30/70 — Given before breakfast and before dinner, target of pre-prandial BG ≤ 100 mg/dl
  Arms: 2

SUMMARY:
To compare efficacy of combination therapy of insulin glargine plus glimepiride and metformin versus 2 injections insulin monotherapy with premixed insulin NPH 30/70 bid in terms of change of HbA1c (baseline to endpoint) to show non-inferiority of insulin glargine plus glimepiride and metformin.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus patients type 2, poorly controlled with oral antidiabetic drug treatment(glimepiride 3 or 4 mg od or any sulfonylurea similar to glimepiride 3 or 4 mg in combination with metformin in a dose at least similar to 850 mg once daily)
* HbA1c value ≥ 7.5 % to ≤ 10.5 %
* FBG ≥ 120 mg/dl (6.6 mmol/l)
* BMI ≤ 35 kg/m²

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2001-12; Primary Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Frequency of subjects with HbA1c ≤ 7.0 % and > 7.0 % | At endpoint

SECONDARY OUTCOMES:
Change of fasting blood glucose | baseline to endpoint
Change of nocturnal & mean daytime blood glucose | baseline to endpoint
Change of fasting plasma glucose | baseline to endpoint and all visits
Frequency of subjects with hypoglycemic events (overall, severe, non-severe, nocturnal, asymptomatic, symptomatic) | Baseline to endpoint
Frequency of hypoglycemic events(overall, severe, non-severe, nocturnal, asymptomatic, symptomatic) | Baseline to endpoint
Frequency of subjects with FBG ≤ 100 mg/dl (5.5 mmol/l), 100 mg/dl < FBG ≤ 120 mg/dl (5.5 mmol/l < FBG ≤ 6.6 mmol/l), 120 mg/dl < FBG ≤ 150 mg/dl (6.6 mmol/l < FBG ≤ 8.3 mmol/l) and > 150 mg/dl (> 8.3 mmol/l) | At endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Christine Kliebe-Frisch, MD, Study Director — Sanofi
Locations (10):
- Sanofi aventis administrative office, Vienna, Austria
- Sanofi-aventis administrative office, Helsinki, Finland
- Sanofi-aventis administrative office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Guildford, United Kingdom